CLINICAL TRIAL: NCT03323099
Title: Using N-of-1 Experiments to Answer Patient Generated Research Questions
Brief Title: Individualized Studies of Triggers of Paroxysmal Atrial Fibrillation
Acronym: I-STOP-AFib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A129075
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation Paroxysmal
MeSH Terms: conditions — Atrial Fibrillation | interventions — Single-Case Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-of-1 (Experimental): Participants in the N-of-1 arm will use the Eureka mobile application and AliveCor device to tracking their AF episode frequency and severity and execute at least one N-of-1 trial with the goal of identifying and better controlling their AF triggers.
  Interventions: Behavioral: N-of-1
- Data Tracking (Placebo Comparator): Participants in the data tracking arm will use the Eureka app and AliveCor device to record daily AF frequency and severity and daily AliveCor readings for a period of 10 weeks.
  Interventions: Behavioral: Data Tracking

INTERVENTIONS:
Behavioral: N-of-1 — Participants in the N-of-1 arm will use the Eureka mobile application and AliveCor device to tracking their AF episode frequency and severity and execute at least one N-of-1 trial with the goal of identifying and better controlling their AF triggers.
  Arms: N-of-1
Behavioral: Data Tracking — Participants in the data tracking arm will use the Eureka app and AliveCor device to record daily AF frequency and severity and daily AliveCor readings for a period of 10 weeks.
  Arms: Data Tracking

SUMMARY:
The I-STOP-Afib study will test the comparative effectiveness of using N-of-1 trials vs. symptom surveillance alone to reduce Atrial Fibrillation (AF) episode frequency and severity and improve quality of life for AF patients. The study will involve randomizing almost 500 paroxysmal AF patients to either AF episode tracking versus engaging in testing the relationship between participant-selected triggers and AF episodes utilizing a mobile-app based N-of-1 study design. Both groups will complete a validated survey to assess AF severity, essentially a measure of quality of life while living with AF, before and after a 3 month testing period.

DETAILED DESCRIPTION:
N-of-1 Trial arm: Participants will use the Eureka mobile application and AliveCor device to execute at least one N-of-1 trial with the goal of identifying and better controlling their AF triggers. Each N-of-1 trial will last a total of 6 weeks and will include up to 3 periods of trigger exposure and 3 periods of trigger elimination with each exposure/elimination period lasting 1 week. Participants will be randomly assigned to start their trial with a period of either trigger exposure or elimination. During each N-of-1 trial, participants will track daily AF duration and severity, daily mood and sleep quality, daily AliveCor tracings and daily trigger exposure. At the end of each trial, participants will be able to review their trial results which will include visualizations of their daily AF symptom and trigger tracking over time. After completing a trial, participants will be instructed to implement any lifestyle changes they deem appropriate based on what they learned from the results of their trial. Participants will implement these changes for a period of 4 weeks during which they will continue to track AF episode duration and severity via the app. At the end of the 4-week lifestyle change period, participants will complete the Atrial Fibrillation Effect on QualiTy of Life survey (AFEQT) and will then have the option of testing another trigger or ending their study participation.

Symptom Surveillance arm: Participants will use the Eureka app and AliveCor device to record daily AF duration and severity, daily AliveCor readings and daily mood and sleep quality for a period of 10 weeks. Participants will be able to visualize their AF, sleep and mood data in real time and will receive a weekly summary of their data via the Eureka app.At the end of the 10-week data tracking period, participants will complete the AFEQT survey and will then have the option of either ending their study participation or crossing over to the N-of-1 trial arm to test their triggers.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic paroxysmal AF
* a smartphone

Exclusion Criteria:

* Non-English speakers
* Children (age < 18 years)
* Patients with plans to substantially change AF management (such as with ablation or change in antiarrhythmic drugs) over the ensuing 6 months
* Unwillingness to test AF triggers.
* Patients who have had an AV node or AV Junction ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Marcus, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcus GM, Modrow MF, Schmid CH, Sigona K, Nah G, Yang J, Chu TC, Joyce S, Gettabecha S, Ogomori K, Yang V, Butcher X, Hills MT, McCall D, Sciarappa K, Sim I, Pletcher MJ, Olgin JE. Individualized Studies of Triggers of Paroxysmal Atrial Fibrillation: The I-STOP-AFib Randomized Clinical Trial. JAMA Cardiol. 2022 Feb 1;7(2):167-174. doi: 10.1001/jamacardio.2021.5010. PMID 34775507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2,987 individuals screened between December 22, 2018 and March 29, 2020, 740 met eligibility criteria, 684 consented, 499 began randomization activities, and 446 completed activities required for implementation of randomization. 320 Participants completed all study activities. The first participant was enrolled March 20th, 2019.
Period: Overall Study
Arm/Group | N-of-1 | Data Tracking
Started | 251 | 248
Completed | 136 | 184
Not Completed | 115 | 64
Not completed — Withdrawal by Subject | 6 | 12
Not completed — Did not complete AFEQT, or failed to start the study period | 109 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-of-1 | Data Tracking | Total
Number analyzed (Participants) | 251 | 248 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.52 (14) | 58.2 (14.04) | 57.85 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 108 | 210
  Male | 149 | 140 | 289
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 8 | 24
  Not Hispanic or Latino | 233 | 233 | 466
  Unknown or Not Reported | 2 | 7 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 9 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 5 | 7
  White | 233 | 228 | 461
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 1 | 4 | 5
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) score [Mean (Standard Deviation); unit: units on a scale] — The Atrial Fibrillation Effect on QualiTy-of-life Questionnaire (AFEQT) evaluates symptoms, daily activities and treatment concerns patients have related to atrial fibrillation (AF or AFib). The AFEQT is the first questionnaire developed and validated for AF patients. Patients score 0 (worst) to 100 (best) Population: 1 participant in the N-of-1 arm had a missing Baseline AFEQT score
  units on a scale
    number analyzed (Participants) | 250 | 248 | 498
    (all) | 74 (19) | 72 (19) | 73 (19)

OUTCOME MEASURES:

1. Primary Outcome: Change in Atrial Fibrillation Effect on QualiTy of Life Survey (AFEQT)
Description: Change in Atrial fibrillation quality of life will be measured by the Atrial Fibrillation Effect on QualiTy of Life survey (AFEQT). The primary outcome will be change in AFEQT score from baseline measurement to measurement at 10 weeks. Change in the AFEQT will compared between the N-of-1 arm and the data tracking arm.
  The Atrial Fibrillation Effect on QualiTy-of-life Questionnaire (AFEQT) evaluates symptoms, daily activities and treatment concerns patients have related to atrial fibrillation (AF or AFib). Patients score 0 (worst) to 100 (best).
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-of-1 | Data Tracking
Number analyzed (Participants) | 135 | 184
units on a scale | 1.7 (13.0) | 0.5 (14.1)

ADVERSE EVENTS:
Time Frame: Data Collected in Primary Data collection period-- over first 10 weeks.
Description: Adverse event information was collected via self report every month-- or twice during the primary data collection period
Arm/Group | N-of-1 | Data Tracking
All-Cause Mortality (participants affected / at risk) | 0/251 | 0/248
Serious Adverse Events (participants affected / at risk) | 8/251 | 16/248
Other Adverse Events (participants affected / at risk) | 0/251 | 0/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-of-1 (N=251) | Data Tracking (N=248)
self report ER visit with AF (Cardiac disorders) | 6 | 9
self report hospital visit with AF (Cardiac disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT03323099/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03323099/SAP_001.pdf